CLINICAL TRIAL: NCT07236619
Title: Durability of Pulmonary Vein Isolation Using a Variable-Loop Biphasic Pulsed Field Ablation Catheter in Patients With Paroxysmal Atrial Fibrillation: a Prospective Remapping Study
Brief Title: Durability of Pulmonary Vein Isolation Using a Variable-Loop Biphasic Pulsed Field Ablation Catheter in Patients With Paroxysmal Atrial Fibrillation
Acronym: VARIFY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Collaborators: Biosense Webster, Inc. (Industry)
Responsible Party: Principal Investigator, Sing-Chien Yap, MD, PhD, Cardiologist-Electrophysiologist, Erasmus Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL-010058
Record Dates: First submitted 2025-11-15; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Paroxysmal AF
Keywords: Varipulse; Catheter ablation; Atrial fibrillation; Paroxysmal atrial fibrillation; Pulmonary vein isolation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- VariPulse treatment group (Experimental): Patients with paroxysmal AF undergoing treatment with the VariPulse catheter
  Interventions: Device: Pulmonary vein isolation with the VariPulse catheter

INTERVENTIONS:
Device: Pulmonary vein isolation with the VariPulse catheter — Pulmonary vein isolation with the VariPulse catheter

SUMMARY:
The VARIFY study is designed to find out how durable pulmonary vein isolation (PVI) is after treatment with the VARIPULSE pulsed field ablation (PFA) system in patients with paroxysmal atrial fibrillation (AF). AF is a common heart rhythm disorder caused by abnormal electrical signals coming from the pulmonary veins. In a PVI procedure, these veins are electrically isolated to prevent AF from recurring. Sometimes, the veins reconnect over time, which can lead to a return of arrhythmia. PFA is a new, non-thermal technology that uses short electrical pulses to safely and precisely treat heart tissue, reducing the risk of damage to nearby structures. The VARIPULSE system is one of these new PFA platforms. In this study, 20 adult patients with paroxysmal AF will undergo PVI using the VARIPULSE system. After 2-3 months, each patient will have a second planned procedure to check whether the pulmonary veins remain isolated. Any reconnections found will be treated immediately. The main goal is to determine how often the pulmonary veins stay durably isolated after the initial VARIPULSE treatment. Secondary goals include assessing the amount of scar tissue in the left atrium, recording any complications, and evaluating rhythm outcomes after one year. The results will help determine how effective and reliable the VARIPULSE system is for long-term treatment of AF.

DETAILED DESCRIPTION:
Rationale: Pulmonary vein isolation (PVI) is the cornerstone of atrial fibrillation (AF) ablation. Pulmonary vein reconnection is associated with recurrence of arrhythmia, thus, durable PVI during the index procedure is important. Recently, pulsed field ablation (PFA) has emerged as a novel nonthermal energy source with high procedural safety and efficacy for PVI. Irreversible electroporation is achieved by the delivery of rapid, high-voltage pulsed electrical fields. Considering differences in catheter design and PFA protocols, it is important to establish PVI durability of the different PFA platforms. In the VARIFY study we will analyze PVI durability of the VARIPULSE platform in patients with paroxysmal AF using a 2-3 months protocol-mandated remapping study regardless of arrhythmia recurrence. Currently, there are no data on PVI durability of the VARIPULSE platform using mandatory remapping. Objective: To assess PVI durability in patients with paroxysmal AF who undergo a firsttime PVI with the VARIPULSE platform. Study design: Prospective, single-center study. Study population: Twenty consecutive adult patients (≥18 years old) with paroxysmal AF who are scheduled to undergo PVI with the VARIPULSE platform. Intervention: Patients will undergo a second invasive procedure 2-3 months after the index PVI. During the second procedure PVI durability will be assessed using high-definition mapping. Any reconnection will be targeted to achieve complete PVI. Main study parameters/endpoints: The primary outcome is the incidence of PV reconnection at the repeat procedure. The secondary outcome include the area of low voltage in the left atrium at the repeat procedure. Nature and extent of the burden and risks associated with participation, benefit, and group relatedness: All patients will undergo a repeat invasive procedure. This second procedure is associated with a similar procedural risk as the first procedure. A potential benefit of a mandated repeat procedure is that early pulmonary vein reconnection is identified and treated. Early treatment of pulmonary vein reconnection is associated with a better arrhythmia outcome.

ELIGIBILITY:
Inclusion Criteria: 1) History of symptomatic paroxysmal AF; 2) Participants who are indicated for a PVI according to the 2020 ESC guidelines for the diagnosis and management of AF; 3) Participants who are willing and capable of undergoing a mandatory repeat procedure 2-3 months after the index procedure; 4) Participants whose age is 18-80 years. 5) Participants who are willing and capable of providing informed consent.

Exclusion Criteria: 1) Any known contraindication to an AF ablation or anticoagulation; 2) History of previous LA ablation or surgical treatment of AF, atrial flutter, or atrial tachycardia; 3) AF secondary to electrolyte imbalance, thyroid disease, or any other reversible or non-cardiac cause; 4) Significant structural heart disease; 5) History of blood clotting or bleeding disease; 6) Severe kidney disease (glomerular filtration rate <30 ml/min/1.73 m2); 7) Stroke or transient ischemic attack <3 months prior to enrollment; 8) Active systemic infection; 9) Pregnant, lactating, or women of childbearing potential who are, or plan to become, pregnant during the time of the study; 10) Participants who are currently enrolled in another investigational study or registry that would directly interfere with the current study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-09-27 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Percentage of pulmonary veins which shows reconnection during the repeat procedure 2-3 months after the index procedure | PV reconnection will be determined in the period from 2 to 3 months after the index procedure.
  During the repeat procedure (2-3 months after the index procedure) the number of pulmonary veins which shows reconnection will be determined. The primary outcome measure is the percentage of pulmonary veins with reconnection.

SECONDARY OUTCOMES:
Extent of low voltage area in the left atrium identified at the repeat procedure 2-3 months after the index procedure | Low voltage area will be determined in the period from 2 to 3 months after the index procedure.
  The low voltage area (<0.5 mV) in the left atrium will be identified during the repeat procedure using high-density 3D-mapping with the OCTARAY catheter.
One-year freedom from atrial arrhythmia after a blanking period of 3 months. | From 3 to 12 months after the index procedure.
  Recurrence of any atrial arrhythmia will be defined as the documentation of atrial arrhythmia on a standard 12-lead ECG or the documentation of ≥30 seconds of atrial arrhythmia on a Holter after a blanking period of 3 months. Twenty-four Holter monitoring will be performed at 6 and 12 months after the ablation procedure.
Percentage of patients with a procedure-related complication | From the index procedure till the 1-year follow-up visit.
  All procedure-related complications will be identified from the index procedure till the 1-year follow-up visit.

CONTACTS AND LOCATIONS:
Overall Officials: Sing-Chien Yap, MD, PhD, Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus MC, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No